CLINICAL TRIAL: NCT05376969
Title: A Multi-center, Open-label, Extension Study to Evaluate the Long Term Safety and Efficacy of DWP16001 add-on to Metformin in Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin
Brief Title: Evaluate the Long Term Safety and Efficacy of DWP16001 add-on to Metformin in Patients With T2DM Inadequately Controlled on Metformin
Acronym: ENHANCE-MEXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001302_Ext
Record Dates: First submitted 2022-01-09; First posted 2022-05-17 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DWP16001 Amg (Experimental): DWP16001 Amg, Tablets, Orally, Once daily
  Interventions: Drug: DWP16001

INTERVENTIONS:
Drug: DWP16001 — DWP16001 Tablets

SUMMARY:
A Multi-center, Open-label, Extension study to Evaluate the long term Safety and Efficacy of DWP16001 add-on to metformin in Patients with type 2 diabetes mellitus inadequately controlled on metformin

ELIGIBILITY:
Inclusion Criteria:

* Participated in the prior phase 3 study (Protocol No: DW_DWP16001302) for meeting the inclusion criteria and completed the study
* Voluntarily decided to participate in the extension study and provided a written consent on the consent form

Exclusion Criteria:

* Withdrawn from the prior phase 3 study (Protocol No: DW_DWP16001302) or expected of having safety issue if taking part in the study in the judgment of the investigator
* Subjects with the following diseases or signs:

  * Diabetic ketoacidosis
  * Moderate to severe renal impairment (estimated glomerular filtration rate [eGFR] < 60 mL/min/1.73 m2
* Females who are pregnant or breast-feeding, or subjects who do not agree to the use of appropriate contraceptive methods throughout the study

Subjects must agree to one of the following appropriate contraceptive methods for subjects or their partners:

① Either surgical sterilization (vasectomy, etc.) or insertion of an intrauterine device (copper loop, intrauterine hormone-containing system), or

② A physical barrier method combined with either systemic hormonal contraceptives or spermicide, or

③ Use of male condom combined with either cervical cap or diaphragm Determined to be ineligible for the study by the investigator, besides the above

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Adverse events (AEs) and adverse events of special interest (AESIs)* at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  *Hypoglycemia, urinary tract infection, genital infection, pollakiuria, or polyuria

SECONDARY OUTCOMES:
Changes from baseline* in HbA1c at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  * Visit 2 (randomization) of the prior phase 3 study (Protocol No: DW_DWP16001302)
Changes from baseline* in FPG at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  * Visit 2 (randomization) of the prior phase 3 study (Protocol No: DW_DWP16001302)
Proportion of subjects achieving HbA1c target of < 7% at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  * Visit 2 (randomization) of the prior phase 3 study (Protocol No: DW_DWP16001302)

CONTACTS AND LOCATIONS:
Locations (1):
- Daewoong pharmatceutical, Seoul, South Korea